CLINICAL TRIAL: NCT00824837
Title: Randomised, Cross Over Pilot Study Comparing Removal of beta2-Microglobulin by Standard Haemodialysis to Haemodialysis With a Novel Dialysis Membrane (P2SH) in Chronic Dialysis Patients
Brief Title: Study of beta2-Microglobulin Removal by Standard Versus New High Cut-Off Haemodialysis Membrane
Acronym: HiCOF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Austin Health (Other Government)
Responsible Party: Rinaldo Bellomo, Austin Health
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 02975; AHHREC02975
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-01

CONDITIONS: Renal Dialysis
Keywords: beta 2 microglobulin; haemodialysis; albumin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): New larger pore membrane
  Interventions: Other: Larger pore haemodialysis membrane; Other: Standard haemodialysis membrane
- B (Active Comparator): Standard haemodialysis membrane
  Interventions: Other: Larger pore haemodialysis membrane; Other: Standard haemodialysis membrane

INTERVENTIONS:
Other: Larger pore haemodialysis membrane — Patients receive haemodialysis sessions 3 times a week. They are randomized to start with either treatment A (experimental arm) or treatment B (active comparator arm) and continue for 2 weeks, followed by a 1-week washout period. The patients then cross-over and receive the other treatment (either B or A) for 2 weeks.
  Other Names: Gambro
Other: Standard haemodialysis membrane — Patients receive haemodialysis sessions 3 times a week. They are randomized to start with either treatment A (experimental arm) or treatment B (active comparator arm) and continue for 2 weeks, followed by a 1-week washout period. The patients then cross-over and receive the other treatment (either B or A) for 2 weeks.

SUMMARY:
The purpose of this study is to determine whether a novel haemodialysis membrane, compared with the standard dialysis membrane, will increase the removal of beta2-microglobulin in chronic dialysis patients.

DETAILED DESCRIPTION:
Despite advances in treatment of kidney diseases, morbidity and mortality of chronic dialysis patients remains unsatisfactory. Standard haemodialysis membranes remove middle-sized molecule solutes poorly such as beta2-microglobulin, which has a pathogenic role in dialysis-related amyloidosis. Pre-dialysis beta2-microglobulin concentration has been shown to be independently predictive of mortality. A new polyamide haemodialysis membrane has been developed with increased pore size to increase the removal of middle-sized uraemic toxins such as beta2-microglobulin. This study aims to evaluate the effectiveness of the new membrane in beta2-microglobulin removal compared with standard haemodialysis membrane in dialysis patients and the degree of increased loss of albumin as a potential limiting factor of its use.

ELIGIBILITY:
Inclusion Criteria:

* Chronic haemodialysis patients for more than 2 years
* Urine output <100 mL per day
* 3 haemodialysis sessions per week
* Permanent arteriovenous dialysis access

Exclusion Criteria:

* Serum albumin <25 g/L

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Beta2-microglobulin removal by new larger pore membrane versus standard haemodialysis membrane | 5 weeks (2 weeks in each arm, 1-week washout period)

SECONDARY OUTCOMES:
Albumin loss with the use of new larger pore membrane compared with standard haemodialysis membrane | 5 weeks (2 weeks in each arm, 1-week washout period)
Removal of low-molecular-weight solutes by new larger pore membrane versus standard haemodialysis membrane | 5 weeks (2 weeks in each arm; 1-week washout period)

CONTACTS AND LOCATIONS:
Overall Officials: Rinaldo Bellomo, MBBS,MD,FRACP, Principal Investigator — Director Intensive Care Research, Austin Health
Locations (1):
- Austin Health, Melbourne, Victoria, Australia